CLINICAL TRIAL: NCT02698644
Title: Hysteroscopic Tubal Occlusion With the Use of Iso Amyl-2-cyanoacrylate
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed I Amer, Professor, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ASU
Record Dates: First submitted 2016-02-19; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Fallopian Tube Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- isoamyl2cyanoacrylate (Experimental): Isoamyl-2-cyanoacrylate will be injected inside fallopian tube hysteroscopically through ureteric catheter
  Interventions: Drug: Isoamyl-2-cyanoacrylate

INTERVENTIONS:
Drug: Isoamyl-2-cyanoacrylate — Isoamyl-2-cyanoacrylate will be injected inside fallopian tube hysteroscopically through ureteric catheter
  Other Names: AMCRYLATE®

SUMMARY:
Is to assess the effectiveness of hysteroscopic tubal application of Iso Amyl-2-cyanoacrylate in occluding uterine tubes of women, which would make it an easy approach for occluding tubes with hydrosalpinx prior to IVF and in tubal sterilization.

DETAILED DESCRIPTION:
The study will be conducted according to the guidelines on human experimentation of the 1975 Declaration of Helsinki. For all patients after taking signed informed consent , transcervical hysteroscopic cannulation of the proximal one centimeter of both fallopian tubes, will be done using a 5 Fr, 42cm long, polyethylene ureteric catheter, where 0.5 ml of Iso Amyl-2-cyanoacrylate (AMCRYLATE®) will be injected in each side.

All the surgical procedures will be performed without anesthesia, only premedication with an NSAID (e.g. NaproxenR) is given orally one hour before the procedure.

Each patient will be under close observation for the first 24 hours postprocedure for any signs of inflammation as abdominal pain, tenderness or fever and for the vital data.

Total abdominal hysterectomy and bilateral salpingoophorectomy will be done, second day, a week, two weeks and three weeks and four weeks after injection,. Hysterectomy samples will be sent to histopathologist to assess the degree of tubal occlusion and the extent and the severity of inflammation in the tubal wall.

ELIGIBILITY:
Inclusion Criteria:

* patients planned for abdominal hysterectomy with well seen tubal ostia through hysteroscope

Exclusion Criteria:

* Any patient with Upper or lower genital tract infection as evidenced by fever, lower abdominal pain or tenderness and abnormal vaginal discharge will be excluded from the study

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
fallopian tube obstruction | from one day to four weeks
  assessed by failure of passage of methylene blue through fallopian tubes after injecting it transcervical in the hysterectomy spacements.

SECONDARY OUTCOMES:
degree and extend of inflammation in the fallopian tubes | from one day to four weeks
  assessments of this outcome will be done by histopathological examination for severity of inflammatory cellular changes and extend of these inflammatory changes through different layers of the wall of the fallopian tubes

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Amer, MD, Principal Investigator — Ain Shams University maternity hospital
Locations (1):
- AIn Shams University Maternity Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided